CLINICAL TRIAL: NCT04357197
Title: Closed-loop Control of Vasopressor Infusion in Critically Ill Patients: A Case Series
Brief Title: Closed-loop Control Mean Arterial Pressure In Intensive Care Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: We did not want to start a case series as we already finished a RCT...SO this study is now outdated
Sponsor: Erasme University Hospital (Other)
Responsible Party: Principal Investigator, Alexandre Joosten, MD PhD, Principal Investigator, Erasme University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P2020-157
Record Dates: First submitted 2020-04-19; First posted 2020-04-22 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Single prospective single center study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Closed-loop (Experimental): Closed-loop administration of norepinephrine in critically ill patients
  Interventions: Device: Closed-loop

INTERVENTIONS:
Device: Closed-loop — The system will be tested to see if it can avoid hypotension

SUMMARY:
The purpose of this case series is to evaluate the performance of a novel closed-loop (automated) vasopressor administration system that delivers norepinephrine using feedback from standard hemodynamic monitor (EV1000 Monitor) from Edwards Lifesciences (IRVINE, USA) in critically ill patients

DETAILED DESCRIPTION:
In this protocol, the investigators will report the percentage of case time in hypotension (defined as Mean arterial pressure (MAP) < 72mmHg) during a two hours study protocol in critically ill patients.

The target MAP will be set at 80 mmHg, and the definition of hypotension is a MAP < 90% of MAP target ( 80 mmHg - 10% = 72 mmHg)

The investigators want to demonstrate that the closed-loop system can prevent hypotension at this specific set point.

The investigators will test the system in a short series of 10-12 critically ill patients in the ICU setting during a two hours study protocol.

Participants will receive standard patient care

Fluids will be given as a baseline crystalloid administration set at 1-2 ml/kg/h

ELIGIBILITY:
Inclusion Criteria:

* All patients in the intensive care unit (awake or under sedation)
* Requiring norepinephrine to maintain a MAP of 80 mmHg
* Equiped with an arterial line

Exclusion Criteria:

* Subjects under 18 years of age
* Subject with Atrial Fibrillation
* Subjects who are pregnant

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-09-25 (Estimated); Primary Completion 2020-12-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of case Time in hypotension (MAP <72 mmHg) | During thetwo hours study protocol
  The primary outcome will be the percentage of case time in predefined MAP target

SECONDARY OUTCOMES:
percentage of case time with MAP >88 mmHg with norepinephrine still running | During the two hours study protocol
  overtreatment
Amount of vasopressors received | During the two hours study protocol
  Amount of vasopressors received (norepinephrine)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Joosten, MD PhD, Principal Investigator — ERASME

IPD SHARING:
Plan to Share IPD: No